CLINICAL TRIAL: NCT02998814
Title: Split Mouth Clinical Trial of Fissure Sealant Retention With Self Etching and Total Etch Bonding Agent
Brief Title: Clinical Follow Up of a Fissure Sealant Placed With Different Adhesive Protocols: 2-Year Randomized Split Mouth Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Bilge Kutuk, Research assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEK 10/13-9
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Fissure Sealant Loss; Caries
Keywords: fissure sealant; etch and rinse; self etch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- acid-etch only (Active Comparator): Selected teeth would receive prophylaxis with pumice using prophylaxis brushes for 20 seconds. The teeth will be isolated with cotton rolls before application of bonding agent. The tooth selected for acid-etch only will be treated with 37% phosphoric acid for 15 seconds followed by rinsing for 30 seconds and then drying with air syringe till frosty white appearance is achieved. Clinpro(3M ESPE) fissure sealant will be applied to pits and fissures and then light cured for 20 seconds.
  Interventions: Other: acid-etch
- self-etch adhesive (Active Comparator): Selected teeth would receive prophylaxis with pumice using prophylaxis brushes for 20 seconds. The teeth will be isolated with cotton rolls before application of bonding agent. The tooth selected for self-etch adhesive will be treated with self-etch adhesive (AdperTM EasyBond, 3M ESPE) for 10 seconds followed by light curing for 20 seconds. Clinpro(3M ESPE) fissure sealant will be applied to pits and fissures and then light cured for 20 seconds.
  Interventions: Other: self-etch adhesive
- etch-and-rinse adhesive (Active Comparator): Selected teeth would receive prophylaxis with pumice using prophylaxis brushes for 20 seconds. The teeth will be isolated with cotton rolls before application of bonding agent. The tooth selected for etch-and-rinse adhesive will be treated with 37% phosphoric acid for 15 seconds followed by rinsing for 30 seconds and then drying with air syringe till frosty white appearance is achieved. Then, etch-and-rinse adhesive (Single BondTM, 3M ESPE) will be treated with for 10 seconds followed by light curing for 20 seconds.Clinpro(3M ESPE) fissure sealant will be applied to pits and fissures and then light cured for 20 seconds.
  Interventions: Other: etch-and-rinse adhesive
- self-etch adhesive after acid-etch (Active Comparator): Selected teeth would receive prophylaxis with pumice using prophylaxis brushes for 20 seconds. The teeth will be isolated with cotton rolls before application of bonding agent. The tooth selected for acid etch + self-etch adhesive will be treated with 37% phosphoric acid for 15 seconds followed by rinsing for 30 seconds and then drying with air syringe till frosty white appearance is achieved. Then, self-etch adhesive (AdperTM EasyBond, 3M ESPE) will be treated with for 10 seconds followed by light curing for 20 seconds.Clinpro(3M ESPE) fissure sealant will be applied to pits and fissures and then light cured for 20 seconds.
  Interventions: Other: self-etch adhesive after acid-etch

INTERVENTIONS:
Other: acid-etch — acid-etch
  Arms: acid-etch only
Other: self-etch adhesive — Self etch (7th generation ) bonding agent
  Other Names: Adper Easy bond 3M ESPE
  Arms: self-etch adhesive
Other: etch-and-rinse adhesive — Total etch bonding agent (5th generation)
  Other Names: Single BondTM, 3M ESPE
  Arms: etch-and-rinse adhesive
Other: self-etch adhesive after acid-etch — acid etch + self-etch adhesive Self etch (7th generation ) bonding agent
  Other Names: acid etch + self-etch adhesive
  Arms: self-etch adhesive after acid-etch

SUMMARY:
The purpose of this study was to evaluate the retention rates of a fissure sealant placed using different adhesive protocols over 24 months.Twenty-four subjects with no restoration and caries received fissure sealants (Clinpro™Sealant, 3M/ESPE) placed with different adhesive protocols. A total of 292 sealants (73 for each group) were placed. The sealants were placed as follows; a-without adhesive (acid-etch only), b-with an etch-and-rinse adhesive (SingleBondTM), c-with a self-etch adhesive (AdperTMEasyBond), d-with acid-etch+self-etch adhesive (AdperTMEasyBond) by two previously calibrated dentists using a table of random numbers. Two other calibrated examiners, independently evaluated the sealants at baseline and at 6-, 12-, 18-, and 24-month recalls. Each sealant was evaluated in terms of caries formation being present or absent and retention using the following criteria: 1=completely retained, 2=partial loss, and 3=total loss. The Pearson χ2 test was used to evaluate differences in retention rates among the sealants for each evaluation period.

DETAILED DESCRIPTION:
Dental caries, which can be encountered by individuals throughout their lives, is one of the most chronic diseases worldwide. Researches have mainly been focusing on the prevention of tooth caries with the awareness of this fact. The use of fluorides as well as pit-and-fissure sealants are the most common preventive applications against caries progression.Modern adhesives combine conventional conditioning, priming and bonding steps (etch-and-rinse adhesives) together into one or two bottle (self-etch adhesives) to ease adhesive protocols. However, it is still suspicious whether modern self-etch adhesives have equal bonding capacity to the conventional etch-and-rinse systems. Therefore, clinical trials are necessary to evaluate long-term adhesive performance of self-etch adhesives compared to the conventional etch-and-rinse ones.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in the current study had good general and oral health and hygiene.
* with no detecatable caries, bruxism, malocclusion, previously placed restorations or sealants on the fissures, or no allergies to resins
* willing to return for follow-up examinations

Exclusion Criteria:

* Third molars
* Uncooperative patients
* Molar teeth with antagonist tooth not present or extracted
* Mentally and physically handicapped patients

Ages: 20 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Changes in retention of sealants from baseline to two years | at baseline and at 6-, 12-, 18-, and 24-month
  The assessment of the retention of sealants (intact, partially lost, completely lost) will be carried out every 6 month for 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: A.Ruya Yazici, DDS, PhD, Study Director — Hacettepe University School of Dentistry
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: pubmed — https://www.ncbi.nlm.nih.gov/pubmed/25864681?dopt=Abstract
- See also: pubmed — https://www.ncbi.nlm.nih.gov/pubmed/11145354?dopt=Abstract